CLINICAL TRIAL: NCT05135611
Title: The Efficacy of the 4-channel Sequential NMES for the Treatment of Sleep Apnea, Single-center Prospective, Open Level, Pilot Study
Brief Title: The Efficacy of the 4-channel Sequential NMES for the Treatment of Sleep Apnea
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Ju Seok Ryu, professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-2112-726-001
Record Dates: First submitted 2021-11-24; First posted 2021-11-26 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 4-channel Sequential NMES (Experimental): After diagnosis of sleep apnea, the registered patient group receives sufficient explanations from the researcher and uses sequential 4-channel electrical stimulation therapy at home, 5 times a week, 60 minutes each, for 8±2 weeks.
  During 4-channel electrical stimulation treatment, study participants kept a treatment log including the number of applications, intensity (mA), and treatment time at home.
  Interventions: Device: 4 channel Electrical Stimulation Device

INTERVENTIONS:
Device: 4 channel Electrical Stimulation Device — electrical stimulation at muscles which related with sleep apnea,. 4-channel NMES is the protocol that provides sequential electrical stimulation to Rt. suprahyoid m (channel 1), Lt.suprahyoid m (channel 2), bilateral thyrohyoid m (channel 3), and biltateral sternothyroid m (channel 4). At this time, channels 1 and 2 start to contract first and stimulate for 1200ms, and channel 3 starts stimulation 150ms after channels 1 and 2, and applies stimulation for 1050ms. Channel 4 starts stimulation 250ms after stimulation of channels 1 and 2 and stimulates it for 950 ms.

SUMMARY:
In the treatment of obstructive sleep apnea, by using sequential 4-channel electrical stimulation treatment, unlike conventional positive pressure devices, it can be done more effectively by improving the strength of the biceps and soft palate, which are the causes of sleep apnea. thought.

DETAILED DESCRIPTION:
Design: Prospective study Inclusion criteria of patient group: Patients aged 19 to 60 years diagnosed with moderate to severe obstructive sleep apnea(n=11) Main outcome measures: AHI (apnea-hypoapnea index), Oxygen saturation lowering variables (minimum oxygen saturation, oxygen saturation time less than 90% (%), oxygen desaturation index (ODI) , REM sleep time and ratio of each). Satisfaction with sleep and discomfort of electrical stimulation treatment before and after treatment were evaluated on the Likert scale.

Evaluate the state of health before and after electrical stimulation treatment through EQ-5D-5L.

ELIGIBILITY:
Inclusion Criteria:

1. Adult males and females between the ages of 19 and 60 who do not fall under the exclusion criteria as study subjects
2. Patients with obstructive sleep apnea syndrome confirmed by polysomnography
3. Those who voluntarily consented to the clinical trial
4. Patients with sleep apnea with moderate or higher apnea hypopnea -

Exclusion Criteria:

1. In case of refusal of inspection
2. Patients who do not agree
3. When instructions cannot be performed due to dementia, mental illness, etc.
4. Patients with sleep apnea due to respiratory failure or cervical spine surgery
5. In case of central nervous system abnormalities such as stroke
6. Pregnant and lactating women
7. Patients who cannot apply the electrical stimulation treatment device due to allergy to electrical stimulation pad (allergic reaction to chemical substances such as silicone, polypropylene, polyethylene, etc.), hypersensitivity reaction, etc.
8. Patients with severe regurgitation during electrical stimulation application
9. Others who have comorbidities (e.g., epilepsy, malignant tumors, severe renal/liver/pulmonary diseases, blood coagulation abnormalities, use of anticoagulants, phlebitis, thermophlebitis, etc.)
10. Those who are judged by other researchers to be unsuitable for this clinical trial (e.g., patients with infectious diseases, those who have inflammation or wounds on the skin at the site of electrical stimulation, and those who believe that electrical stimulation can cause abnormalities in the body regardless of disease) judged person)
11. Those who have been diagnosed with a disease that cannot be stimulated

    i. In patients with peripheral neuropathy (ex. Guillain-Barré syndrome), the electric stimulator does not induce muscle contraction, so it is ineffective.

    ii. Patients with congenital myopathy and amyotrophic lateral sclerosis do not receive help because muscle contraction is not induced.
12. Patients with sleep apnea due to pharyngeal muscle weakness or abnormal muscle contraction pattern
13. Persons with pacemakers and other internal electrical stimulators
14. Patients with a history of surgery in the area where the medical device is applied, or in the upper respiratory tract or surrounding area
15. Structural diseases such as 'tonsil hypertrophy' and 'soft palate' that can cause 'obstructive sleep apnea' (examined by physical examination)

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 11 (Estimated)
Dates: Start 2022-07-05 (Actual); Primary Completion 2022-10-14 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
The difference value of polysomnography before and after treatment | After 8±2 weeks of treatment at home, it is performed within 2 weeks of the end of treatment.
  The index for primary efficacy evaluation is the apnea hypopnea index (AHI) calculated based on polysomnography.

SECONDARY OUTCOMES:
Sleep satisfaction and discomfort | After 8±2 weeks of treatment at home, it is performed within 2 weeks of the end of treatment.
  Satisfaction and discomfort during sleep before and after treatment are evaluated using the Likert Scale scale and verified using the EQ-5D-DL questionnaire that evaluates each individual's health status in a self-written method.

CONTACTS AND LOCATIONS:
Overall Officials: InYoung Yoon, M.D, PhD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Department of Rehabilitation Medicine, Seoul National University Bundang Hospital, Seoul National University College of Medicine, Seongnam-si, Gyeonggi-do, South Korea